CLINICAL TRIAL: NCT06087484
Title: The Effect of Mindfulness Intervention for Emotional Distress of Insomnia People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20230922
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Emotional Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIED-I group (Experimental): Provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and sleep problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress and Insomnia (MIED-I)
- Waitlist control group (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress and Insomnia (MIED-I) — The MIED-I program integrates the rationales and practices from the Unified Protocol for Treatment of Emotional Disorders (UP) and Mindfulness based Interventions. Formal mindfulness exercises (e.g., body scan, mindful breathing, and mindful stretching) and informal mindfulness practices (e.g., mindful tooth brushing) were adapted from Mindfulness based intervention (MBIs).Also, a portion of the CBT-I will be added to the course to provide psychoeducation for insomnia. Variables that have been shown to be effective in interventions for insomnia in past studies, such as awareness, non-responsiveness, and self-compassion, will also be added to better alleviate insomnia symptoms
  Arms: MIED-I group

SUMMARY:
Exploring the Effectiveness of a mindfulness intervention for Insomniacs with Emotional Distress Comparing the intervention effects of two mindfulness interventions

DETAILED DESCRIPTION:
Insomnia is a term used to refer to "not sleeping well," which can include difficulty falling asleep at night, excessive dreaming, frequent awakenings that make it difficult to fall asleep, waking up too early, and other symptoms of dissatisfaction with the length and quality of sleep. Some scholars believe that insomnia also belongs to a type of emotional disorder. Although few studies have been able to definitively describe insomniacs' responses to negative emotions, insomniacs inhibit or avoid efforts to suppress emotional experiences in relation to sleep disorders, and insomnia has been associated with the use of sleep-related safety behaviors, which are a form of avoidant coping that maintains symptoms by reinforcing maladaptive belief. Also, 40% of insomniacs have comorbid psychiatric disorders. Longitudinal studies have shown that anxiety and depression present with sleep problems are more severe and also increase the risk of illness. Thus, the relationship between sleep problems and anxiety and depression may be bidirectional. For example, the close association between insomnia and depression may be due to the fact that sleep and mood regulation share underlying pathophysiological mechanisms, and there may be some neuroendocrine similarities between insomnia and depression. All of this evidence suggests that insomnia and comorbid psychiatric disorders can lead to a vicious cycle of reciprocal causation and, at the same time, are likely to respond to the same therapeutic interventions. In such a context, SCT, SRT, and CBT-I therapies that solely target insomnia symptoms may not bring more benefits to patients beyond insomnia symptom relief and do not address the cycle between insomnia and anxiety and depression. Therefore, the development and availability of alternative treatment modalities can improve insomnia patients' access to psychotherapy, as well as the overall efficiency of treatment.

There is now a large body of evidence that various forms of positive mindfulness-based interventions can be effective in improving sleep quality and alleviating insomnia symptoms, and can thus be an adjunct to sleep therapy, but there is still room for improvement. The original positive thought-based intervention programs for insomnia, such as MBSR, MBCT, and MBT-I, are all conducted offline, etc., and are susceptible to a variety of additional factors. As an emerging intervention program for insomnia, the number of therapists who can master MBT-I is even more limited.

There is preliminary evidence that the MIED (Mindfulness Intervention for Emotional Disturbance) program has shown significant improvements in the mental health of patients with anxiety and depression. Meanwhile, if investigators follow the above scholars' analysis of insomnia, which is also a type of emotional disorder, then through the MIED program, participants can relieve both anxiety and depression and insomnia, which is more cost-effective than the previous program that only focuses on insomnia. which is more cost-effective than the previous positive thinking intervention program for insomnia only.

This study proposes to develop a special version of the original MIED program, the Mindfulness Intervention for Emotional Distress and Insomnia (MIED-I). Adding part of the original CBT-I, the gold standard for insomnia treatment, this part of the adjustment will be mainly reflected in the psycho-education for insomnia, while keeping the basic framework of the original four strategies of MIED and the corresponding explanations and exercises unchanged, but at the same time, more directly to solve the main insomnia disturbances.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with scores greater than 21 on the Kessler Psychological Distress Scale, and Pittsburgh sleep quality index scores greater than 5, Insomnia severity index's scores greater than 8

Exclusion Criteria:

* Subjects who have participated in mindfulness-based projects (especially MIED), and/or the current frequency of meditation practice is more than once a week; Patients with schizophrenia or psychotic affective disorder, current organic; mental disorder, substance abuse disorder, and generalized developmental disorder; Subjects at risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-16 (Estimated); Primary Completion 2024-01-23 (Estimated); Study Completion 2024-01-28 (Estimated)

PRIMARY OUTCOMES:
Changes of Five Facet Mindfulness Questionnaire-short form during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Weekly changes of 10-item Kessler Psychological Distress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress
Weekly changes of Overall Anxiety Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
. Weekly changes of Overall Depression Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Weekly changes of Insomnia severity index during the intervention | pre-intervention; after the 3rd week intervention; after the 7-week intervention; one month after intervention
  The ISI is a self-report scale used to detect the severity of insomnia, with scores ranging from 0 to 28; the higher the score, the more severe the insomnia.
Weekly changes of Pittsburgh sleep quality index during the intervention | pre-intervention; after the 3rd week intervention; after the 7-week intervention;one month after intervention
  The Pittsburgh Sleep Index is a self-measured scale used to measure the quality of sleep over the past month, higher the score, the poorer the quality of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No